CLINICAL TRIAL: NCT00150982
Title: In Vivo Induction of T Cell Apoptosis by Alefacept (LFA-3/IgG1 Fusion Protein, Amevive) in Patients With Psoriasis: An Investigator-Initiated, Open-Label, Mechanism of Action Study
Brief Title: Alefacept Mechanism of Action in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Biogen (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4588
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Psoriasis
Keywords: psoriasis; alefacept
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mechanism of action of alefacept

SUMMARY:
To determine the mechanism of action of alefacept in patients with psoriasis.

DETAILED DESCRIPTION:
The purpose of the study is to better understand the mechanism of action of an FDA approved drug (alefacept). Subjects enrolled will be given alefacept 7.5 mg intravenously on a weekly basis for 12 weeks. Response is assessed by improvement in the PASI score. The responders will get no further treatment and the nonresponders will receive additional 4 weeks of therapy. Skin biopsies will be obtained throughout the study and T-cell apoptosis will be correlated to clinical response. There is no placebo group. The duration of the study is approximately 1 year.

ELIGIBILITY:
Inclusion Criteria

* Alefacept is indicated for the treatment of adult patients (18 years or older) with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy. Patients must have at least one plaque of least 2.5 cm in diameter (for biopsies).

Exclusion Criteria

* CD4 < 400/ml
* WBC less than lower level of normal for the reporting laboratory
* < 5% Body Surface Area involved with psoriasis
* Serious infection e.g., latent or active tuberculosis
* History of AIDS or Hepatitis B,C, all internal cancers, lymphoma, untreated cutaneous basal or squamous cell carcinoma
* Systemic anti-psoriasis medications and phototherapy within 28 days of the first dose of Alefacept
* Topical anti-psoriasis medications within 14 days of the first dose of Alefacept, except for moisturizers, tar shampoos (exception, Elidel is permitted to be applied on the face, groin and axillae areas. These areas are not biopsied.)
* Inability to understand consent form or comply with study requirements
* Pregnancy or lactation
* Concurrent medical illness that would make participation in this clinical trial ill-advised
* Any contraindications to using alefacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9
Dates: Start 2003-09; Study Completion 2005-02

PRIMARY OUTCOMES:
To determine if alefacept induces apoptosis in circulating T cells and plaque T cells in psoriasis patients in vivo

SECONDARY OUTCOMES:
To determine if apoptosis of circulating or plaque T cells in vivo is a better predictor of clinical response than are circulating CD4 T cell counts.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gottlieb, MD, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ Clinical Research Center, New Brunswick, New Jersey, United States